CLINICAL TRIAL: NCT05427409
Title: Ingestion of Beta-alanine Improves Neuromuscular Performance in Well-trained Tennis. A Randomized Controlled Trial.
Brief Title: Ingestion of Beta-alanine Effects in Well-trained Tennis Players
Acronym: BETA_TENNIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: University of Seville (Other); University of Greenwich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UFran_Vitoria
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Beta-alanine; Placebo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-alanine supplementation (Active Comparator): Beta-alanine (4.8 grams) pills (Crown Nutrition, Haro, Spain) in four doses each day during a 4-week supplementation period.
  Interventions: Dietary Supplement: Beta-alanine supplementation
- Placebo supplementation (Placebo Comparator): Placebo (4.8 grams) pills (Crown Nutrition, Haro, Spain) contain fructose (300mg) and excipients (1200 mg) such as cellulose, calcium phosphate, silicon dioxide and magnesium stearate in four doses each day during a 4-week supplementation period.
  Interventions: Dietary Supplement: Beta-alanine supplementation

INTERVENTIONS:
Dietary Supplement: Beta-alanine supplementation — In a randomized order, two groups (n=7) was randomly assigned to beta-alanine and placebo during a 4-weeks period
  Other Names: Placebo supplementation

SUMMARY:
Beta-alanine is considered as ergogenic aids with good to strong evidence for improving sports performance in specific sports context scenarios. However, most of the studies has been realized in endurance, with limited evidence in intermittent sports, especially in racket sports. Thus, the aim of this study was to explore the effects of 4-weeks ingestion of beta-alanine on neuromuscular performance in well-trained tennis players.

DETAILED DESCRIPTION:
Fourteen tennis players (23.3 ±3.7 years) between 50-250 national tennis ranking participated in this study. Participants were randomly divided into two groups that realized a neuromuscular battery after beta-alanine (4.8 gr/daily during 4-weeks) or placebo (i.e., fructose) (4.8 grams/daily during 4-weeks). Before and after the supplementation period tennis performed a neuromuscular test battery in a tennis court consisted in different test such as; serve velocity, countermovement jump, isometric handgrip strength, 10-m sprint, modified 5-0-5 agility test and repeated sprint ability. After 48 h of the realization of neuromuscular test battery, tennis players performed VO2max consumption test (i.e., treadmill).

ELIGIBILITY:
Inclusion Criteria:

* Well-trained tennis players, between 18-35 years old (50-200 between tennis ranking)

Exclusion Criteria:

* Suffering from any chronic pathology or an injury in the month prior to the investigation.
* Intolerance to beta-alanine ingestion
* Amateur tennis players.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Repeated sprint ability test. | 4-weeks
  Infrared photocells system (Microgate, Italy)
VO2 max treadmill test | 4-weeks
  Using VO2 max analyzer (Ergostik, Geratherm Respiratory, Ergostik, Geratherm, Germany)

SECONDARY OUTCOMES:
Serve velocity | 4-weeks
  Stroke velocity radar gun (Radar Pocket, South Korea)
Contermovement Jump | 4-weeks
  Contact Jump (Chronojump, Spain)
10m sprint | 4-weeks
  Infrared photocells system (Microgate, Italy)
Isometric handgrip strength | 4-weeks
  Hand held dynamometer (Takei, Japan)
Modified agility test 5-0-5 | 4-weeks
  Infrared photocells system (Microgate, Italy)

CONTACTS AND LOCATIONS:
Overall Officials: Iñaki Quintana García-Milla, PhD, Principal Investigator — Universidad Francisco de Vitoria
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No